CLINICAL TRIAL: NCT03176706
Title: Assessment of Dried Blood Spot Thyroglobulin in Pregnant Women to Redefine the Range of Median Urinary Iodine Concentration That Indicates Adequate Iodine Intake
Brief Title: Assessment of Dried Blood Spot Thyroglobulin and Urinary Iodine Concentration in Pregnant Women
Acronym: STRIPE
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr., Swiss Federal Institute of Technology
Other Study IDs: STRIPE
Record Dates: First submitted 2017-06-02; First posted 2017-06-05 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Iodine Deficiency; Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Lebanese pregnant women: Pregnant women which are suspected to have mild to moderate iodine deficiency but are otherwise health and living in the Lebanon.
  Interventions: Other: no intervention
- Thai pregnant women: Pregnant women which are suspected to have mild to moderate iodine deficiency but are otherwise health and living in Thailand.
  Interventions: Other: no intervention
- South African pregnant women: Pregnant women which are suspected to have mild to moderate iodine deficiency but are otherwise health and living in South Africa.
  Interventions: Other: no intervention
- New Zealand pregnant women: Pregnant women which are suspected to have mild to moderate iodine deficiency but are otherwise health and living in New Zealand.
  Interventions: Other: no intervention
- Swedish Pregnant women: Pregnant women which are suspected to have mild to moderate iodine deficiency but are otherwise health and living in Sweden.
  Interventions: Other: no intervention
- Peruvian pregnant women: Pregnant women which are suspected to have mild to moderate iodine deficiency but are otherwise health and living in Peru.
  Interventions: Other: no intervention
- Russian pregnant women: Pregnant women which are suspected to have mild to moderate iodine deficiency but are otherwise health and living in Russia.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this is a completely observational study, NO INTERVENTION

SUMMARY:
To avoid iodine deficiency and its consequences in pregnant women and their offspring, women should reach a sufficient iodine intake long before conception. To monitor iodine status, median urinary iodine concentration (UIC) is widely used in pregnant women (PW). Thyroglobulin (Tg) us another marker used to assess iodine status . In this study, urine samples as well as dried blood spots will be collected to measure UIC and Tg (as well as other hormones to define thyroid function) in PW. The results shall be used to reassess the threshold which defines iodine status in PW according to UIC.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy
2. No major medical illness, no thyroid disease, and taking no chronic medication
3. No use of iodine containing dietary supplements
4. No use of iodine-containing X-ray /CT contrast agent or iodine containing medication within the last year
5. Aged between 18 and 44 at enrollment
6. Singleton pregnancy
7. Non-smoking
8. Residence at study site since 12 months or longer

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women aged from 18 to 44 years, living since 12 months or longer in the respective country.
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration and Thyroglobulin concentration in pregnant women. | June 2018
  Analysis of urine and blood samples to find urinary iodine concentration and Thyroglobulin concentration of each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Otago, Dunedin, Otago, New Zealand